CLINICAL TRIAL: NCT07276477
Title: Effects of Inspiratory Muscle Training Via a Mobile Respiratory Trainer (AiroFit PRO™) on Pulmonary Function, Muscle Strength, and Quality of Life in Hemiplegic Individuals: A Randomized Controlled Study
Brief Title: Inspiratory Muscle Training After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Ali Yavuz Karahan, Professor, Uşak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ayk & Stroke
Record Dates: First submitted 2025-11-28; First posted 2025-12-11 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Exercise; Pulmonary
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Intervention Model Description: A prospective, single-blind (assessor-blinded), two-arm, randomized controlled trial with a 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Masking Description: In this randomized controlled trial, assessor blinding (also known as single-blinding) refers to the practice where the healthcare professionals responsible for measuring the study's primary and secondary outcomes are kept unaware of which intervention group (AiroFit™ PRO or Pursed-Lips Breathing) each participant has been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device-Guided Inspiratory Muscle Training (AiroFit™ PRO) (Experimental): * Device: The AiroFit™ PRO mobile respiratory trainer will be used.
  * Principle: The device provides adjustable, pressurized resistance to inhalation and exhalation, with real-time visual feedback provided via a connected smartphone application.
  * Procedure:
    1. Participants will be seated in a comfortable chair.
    2. The initial training intensity (resistance level) will be set based on the device's calibration feature, which typically starts at 50-60% of the individual's maximal inspiratory pressure (MIP).
    3. Participants will be instructed to perform slow, deep inspirations through the device, following the visual pacing and targets on the smartphone app.
    4. The training protocol will consist of structured breathing exercises as per the AiroFit™ PRO's built-in programs, which include cycles of inspiratory load, breath-holds, and expiratory phases.
  Interventions: Other: Device-Guided Inspiratory Muscle Training; Other: Concomitant Care
- Pursed-Lips Breathing Training (Active Comparator): * Device: None. This is a non-device, technique-based breathing exercise.
  * Principle: Pursed-Lips Breathing (PLB) is a simple breathing technique that involves inhaling through the nose and exhaling slowly and gently through pursed lips, creating back-pressure to keep small airways open.
    * Procedure:
      1. Participants will be seated in a comfortable chair with their shoulders relaxed.
      2. They will be instructed by the physiotherapist to:
         1. Inhale slowly and deeply through the nose for a count of 2 seconds.
         2. Pucker their lips as if to whistle.
         3. Exhale slowly and gently through the pursed lips for a count of 4 seconds (aiming for an I:E ratio of 1:2).
      3. The session will consist of continuous cycles of this breathing pattern for the full 15-minute duration.
      4. The physiotherapist will provide verbal cues and correction to ensure proper technique throughout the session.
  Interventions: Other: Pursed-Lips Breathing Training; Other: Concomitant Care

INTERVENTIONS:
Other: Device-Guided Inspiratory Muscle Training — The AiroFit™ PRO mobile respiratory trainer will be used.
  Arms: Device-Guided Inspiratory Muscle Training (AiroFit™ PRO)
Other: Pursed-Lips Breathing Training — Technique-based breathing exercise
  Arms: Pursed-Lips Breathing Training
Other: Concomitant Care — All participants will continue to receive their standard conventional neurorehabilitation therapy (e.g., physiotherapy, occupational therapy) as prescribed by their physician. This concomitant care will be documented for both groups to ensure equivalence.

SUMMARY:
Objective: To investigate and compare the efficacy of a 6-week, supervised respiratory training program using the AiroFit PRO™ mobile respiratory trainer against traditional Pursed-Lips Breathing exercises in individuals with hemiplegia.

Study Design: A single-blind, two-arm, randomized controlled trial.

Participants: Ambulatory adults with stable hemiplegia (≥3 months post-stroke), who are medically stable and able to follow commands.

Interventions: Participants will be randomly assigned to one of two groups:

Experimental Group: Will perform Inspiratory Muscle Training using the AiroFit PRO™ device for 15 minutes/day, 5 days/week, for 6 weeks. The intensity will be progressively increased.

Active Control Group: Will perform Pursed-Lips Breathing exercises for an identical duration and frequency.

Primary Outcomes: Changes in pulmonary function tests, including Forced Vital Capacity (FVC), Forced Expiratory Volume in 1 second (FEV1), and Maximal Inspiratory Pressure (MIP).

Significance: This study will provide high-level evidence on the utility of smart, device-guided respiratory training as a novel component of neurorehabilitation, potentially offering a more effective strategy to improve respiratory health and overall recovery in hemiplegic patients compared to standard breathing exercises.

DETAILED DESCRIPTION:
Hemiplegia, a cardinal feature of post-stroke morbidity, is characterized by unilateral motor weakness and paralysis, leading to profound physical deconditioning. While rehabilitation efforts have traditionally focused on limb function and ambulation, the critical role of respiratory muscle strength in overall functional capacity and quality of life is increasingly recognized. Individuals with hemiplegia frequently exhibit diaphragmatic weakness and impaired pulmonary function on the affected side, a condition often termed "respiratory hemiplegia." This can result in restrictive lung patterns, reduced cough efficacy, and increased susceptibility to respiratory complications, further diminishing physical performance and independence.

Inspiratory Muscle Training (IMT) has emerged as a targeted intervention to address this deficit. By providing resistance during inhalation, IMT aims to strengthen the diaphragm and accessory respiratory muscles, analogous to strength training for limb muscles. Conventional IMT has shown promise in various populations; however, its application in hemiplegia can be limited by a lack of motivation, difficulty with handling devices, and the absence of biofeedback.

The advent of smart, mobile respiratory trainers, like the AiroFit PRO™, offers a potential solution to these limitations. These devices provide real-time visual feedback and structured training programs, which may enhance patient engagement, ensure correct technique, and allow for precise progression of training intensity. While the benefits of standard IMT are being explored, the specific efficacy of this new generation of technologically assisted devices in a hemiplegic population remains insufficiently investigated.

Therefore, this study is designed to bridge this gap in clinical knowledge. We hypothesize that a structured IMT program using the mobile AiroFit PRO™ device will lead to significant improvements in respiratory muscle strength, pulmonary function parameters, and overall quality of life in individuals with hemiplegia compared to a control group.

Participants: Ambulatory adults with stable hemiplegia (≥3 months post-stroke), who are medically stable and able to follow commands.

Interventions: Participants will be randomly assigned to one of two groups:

Experimental Group: Will perform Inspiratory Muscle Training using the AiroFit PRO™ device for 15 minutes/day, 5 days/week, for 6 weeks. The intensity will be progressively increased.

Active Control Group: Will perform Pursed-Lips Breathing exercises for an identical duration and frequency.

Primary Outcomes: Changes in pulmonary function tests, including Forced Vital Capacity (FVC), Forced Expiratory Volume in 1 second (FEV1), and Maximal Inspiratory Pressure (MIP).

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis: A confirmed diagnosis of unilateral hemiplegia or hemiparesis (e.g., secondary to ischemic or hemorrhagic stroke), sustained at least 3 months prior to enrollment.
* Age: Aged between 18 and 80 years.
* Stable Medical Condition: Medically stable, as determined by the treating physician, with no changes in their primary rehabilitation regimen or medication for spasticity/neurological condition in the past 4 weeks.
* Cognitive & Communication Ability: Sufficient cognitive function and language comprehension to understand and follow simple commands and provide informed consent, as assessed by a Mini-Mental State Examination (MMSE) score of ≥ 24 (or a similar validated tool).
* Respiratory Status: Able to perform forced expiratory maneuvers for spirometry and tolerate the breathing training protocols.

Exclusion Criteria:

* Pre-existing, significant respiratory diseases (e.g., severe COPD, asthma, pulmonary fibrosis, active lung cancer).
* Unstable cardiovascular conditions (e.g., uncontrolled hypertension, unstable angina, recent myocardial infarction within the past 6 months, congestive heart failure NYHA Class III or IV).
* Inability to achieve a proper seal with the breathing trainer mouthpiece due to facial muscle weakness or other anatomical reasons.
* Inability to commit to the 6-week training and assessment schedule

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-05-11 (Estimated); Study Completion 2026-06-11 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | T0: baseline (pre-intervention) / T1: post-intervention (after 6 weeks)
  The maximum volume of air, in liters, that a participant can forcibly and completely exhale after taking the deepest possible breath. It reflects the overall function and size of the lungs.
Forced Expiratory Volume in 1 second (FEV1) | T0: baseline (pre-intervention) / T1: post-intervention (after 6 weeks)
  The maximum volume of air, in liters, that a participant can forcibly exhale in the first second of the FVC maneuver. It is a key indicator of airway obstruction.
FEV1/FVC Ratio | T0: baseline (pre-intervention) / T1: post-intervention (after 6 weeks)
  The ratio of FEV1 to FVC, expressed as a percentage. This is the primary index used to diagnose and categorize the presence and severity of obstructive lung defects. A reduced value indicates airflow limitation
Forced Expiratory Flow 25-75% (FEF25-75) | T0: baseline (pre-intervention) / T1: post-intervention (after 6 weeks)
  The average rate of airflow, in liters/second, during the middle half (25% to 75%) of the FVC maneuver. It is considered a sensitive measure of airflow in the smaller peripheral airways.

SECONDARY OUTCOMES:
The Six-Minute Walk Test | T0: baseline (pre-intervention) / T1: post-intervention (after 6 weeks)
  The Six-Minute Walk Test (6MWT) is a functional walking test in which the distance that a client can walk within six minutes is evaluated. This test has been used to assess individuals with stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Buker, Professor, Study Director — Pamukkale University
Locations (1):
- University of Usak, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The IPD and supporting documents will not be made available until the study has been published.